CLINICAL TRIAL: NCT06486935
Title: City For All Ages: Elderly-friendly City Services for Active and Healthy Ageing
Status: Recruiting | Type: Observational
Sponsor: National University of Singapore (Other)
Collaborators: University of Sfax (Other)
Responsible Party: Principal Investigator, Oteng Ntsweng, Clinical Assistant Professor, Arizona State University
Other Study IDs: SACIoTStudy
Record Dates: First submitted 2024-02-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Baseline/Control Phase; Intervention Phase

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Time period prior to & after the implementation of IoT sensors: Since our study involves a single group of 19 participants, we will evaluate their quality of life at two different times: before and after the introduction of IoT sensors.
  Interventions: Device: IoT sensors; Other: Traditional/Manual elderly monitoring

INTERVENTIONS:
Device: IoT sensors — The proposed assistive Activities of Daily Living (ADL) monitoring system consists of ambient infrared sensors embedded seamlessly into the living environment, and a visualization app. Multimodality sensors with wireless data transmission capability will be installed at different locations (e.g. bedroom, kitchen, toilet, bathroom, living room, etc.) to monitor and detect the activities performed by individual elderly, such as cooking, sleeping, going to the bathroom, going out of the apartment or potential wandering, bathroom falls, etc. In addition, a micro-bend fiber optic pressure sensor mat will be placed unobtrusively below the bed mattress to measure the elderly's heart and respiratory rates during sleep. This mat helps provide information on the quality of sleep and sleep-wake rhythms of the elderly with sleep disorders. The collected data will then be transferred through a secured gateway with Raspberry Pi to a dedicated server for data processing and analysis.
Other: Traditional/Manual elderly monitoring — Traditional elderly care without the use of IoT sensors.

SUMMARY:
Many city-dwelling elderly people can be greatly affected after a minor change in their living or health conditions. Mild Cognitive Impairment (MCI), early dementia and frailty are among the most common risks with deep consequences on elderly's and caregivers' quality of life. Through the new wave of Information and Communication Technologies (ICT), Internet of Things (IoT) and smart city system, it is now possible to help individuals capture and make use of their personal data in a way that will help them maintain their independence for longer. The City for all Ages project will create an innovative service based on:

* ICT-enhanced early detection of risk related to frailty
* ICT-enhanced interventions that can help the elderly population to improve their daily life and also promote positive behaviour change

Through real-life pilot sites in Singapore in collaboration with TOUCH Senior Activity Centre (SAC) and the Housing Development Board (HDB), this project explores how data on individual behaviours captured through indoor and outdoor sensors could be used for the observation and detection of the following parameters:

* Activity of Daily Living (ADL): nutrition, hygiene, sleep activity
* Mobility: physical activity, going-out frequency and length
* Cognition: forgetfulness, early signs of mental decline
* Socialization: senior activity centre visits, activities attended, other places of interests visits

This 2-year project comprises of 3 phrases involving 10 healthy elderly living in HDB home in phases 1 and 2 and 100 elderly in phase 3. Our focus is to use sensing technologies installed in the elderly's home to monitor and detect their activities of daily living. Sensor data that is collected will then be analyzed to identify relevant behaviours of individuals, and to detect behavioral changes that can be correlated with risks of MCI/frailty. The appropriate ICT based interventions (e.g. data visualization and alerts to caregivers) will then be applied to mitigate these risks. Additionally, psychosocial data related to the elderly's quality of life, social activity participation and activities of daily living will also be collected via interviews and activity logs to evaluate the outcomes of our technology intervention.

DETAILED DESCRIPTION:
Like many developed countries, Singapore faces the challenges of an ageing population. The number of Singaporeans aged 65 and above is increasing rapidly as population growth slows. The number of seniors has doubled from 220,000 in 2000 to 440,000 in 2015, and is expected to increase to 900,000 by 2030. Amongst the elderly people, close to 10% are living alone (from 35,000 in 2012 to 83,000 by 2030). The changing demographic not only increases healthcare costs but also the demand on healthcare services and care provision.

Preventing frailty and MCI is key for the elderly to maintain their day-to-day activities and remain healthy and independent at home. Prior research has shown that frailty, like disability, is a dynamic process with older individuals moving back and forth between different frailty states. Transition to frailty is a gradual progression that occurs over the course of several months or years, and there are surprisingly high rates of recovery. However, it is important to intervene within the right time window before a person goes into full blown frailty. Hence it is important to detect the onset and progression of frailty and to identify the factors that may facilitate transitions to less frail states. This can inform the development of interventions to manage elderly at risk for fraility.

City for All Ages project seeks to demonstrate that smart cities can play a pivotal role in "prevention" (i.e. the early detection and consequent intervention) of MCI and frailty-related risks. The core idea is that "smart cities", enabled by the deployment of sensor technologies and analytics can collect data about individuals: a) to identify segments of population potentially at risk, in order to start more stringent monitoring; b) to closely monitor selected individuals, in order to start a proactive intervention. In both cases adverse changes of behaviors that are identified through a set of indicators can prompt preventive actions. The aim is to advance the research on healthcare towards a proactive rather than reactive system.

The research team will leverage the existing experimentations and pilot sites that have focused on detection of elderly risky behaviors both in France and Singapore. Lessons learnt from dealing with challenges either in terms of understanding the data (such as false positives, meaningful information, etc.) or providing the appropriate and timely intervention (such as difficulty in identifying and organizing the intervention effectively, large panel of stakeholders, excessive solicitation of caregivers, etc.) would be useful for this project.

Our goal is to use sensing technologies installed in the elderly's home to monitor and detect their activities such as cooking, sleeping, going to the bathroom, going out of the apartment or potential wandering, bathroom falls. Sensor data will be collected unobtrusively and managed using a privacy-aware linked open data paradigm. Basic reasoning and learning algorithms will be applied to the data to identify relevant behaviours of individuals, and to detect behavioral changes that can be correlated with risks of MCI/frailty. The appropriate ICT based interventions (e.g. data visualization and alerts to caregivers) will then be applied to mitigate these risks.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively abled elderly people-as determined by the senior activity center staff during the identification of potential participants.
* Living alone or with no more than 2 flatmates
* Resident of an HDB apartment
* Preferably, apartments with WIFI internet connection
* English or Chinese speaker-in phase 1, only mandarin speakers will be included in the study. Depending on the number of dialect speaking elderly in the residences, in subsequence phases, dialect speaking subjects will be included.
* Member of the Senior Activity Centre
* Agree to share their activity of daily living (ADL) data with the research team, the Senior Activity Centre team and (if applicable) their designated relatives

Exclusion Criteria:

* Those who don't meet the aforementioned inclusion criteria
* Have Severe disabilities
* Have reduced mobility (using wheelchair)
* Have severe dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Below are the inclusion criteria for elderly participants:
  * Cognitively abled elderly people-as determined by the caregivers.
  * Living alone or with no more than 2 flatmates
  * Resident of an HDB apartment
  * Preferably, apartments with WIFI internet connection
  * English or Chinese speaker-in phase 1, only mandarin speakers will be included in the study. Depending on the number of dialect speaking elderly in the residences, in subsequence phases, dialect speaking subjects will be included.
  * Member of the Senior Activity Centre
  * Agree to share their activity of daily living (ADL) data with the research team, the Senior Activity Centre team and (if applicable) their designated relatives
  * English or Chinese speaker
  * Have a smartphone, tablet or a computer
Sampling Method: Non-Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2016-01-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Elderly's Perceived Quality of Life at 6 Months | 6 months
  The older adults' perceived quality of life reported during semi-structured interviews

SECONDARY OUTCOMES:
Change from Baseline in the Caregiver's Perceived Fatigue at 6 Months | 6 months
  Caregivers' perceived fatigue levels reported during semi-structured interviews

CONTACTS AND LOCATIONS:
Locations (2):
- Institut Mines Télécom (IMT), Paris, France
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to ethical reasons, we cannot share IPD. Only aggregated results will be shared in a publication.

REFERENCES:
- [Derived] Ntsweng O, Kodys M, Ong ZQ, Zhou F, Marasse-Enouf A, Sadek I, Aloulou H, Tan SS, Mokhtari M. Lessons Learned From the Integration of Ambient Assisted Living Technologies in Older Adults' Care: Longitudinal Mixed Methods Study. JMIR Rehabil Assist Technol. 2025 Jun 11;12:e57989. doi: 10.2196/57989. PMID 40369868